CLINICAL TRIAL: NCT06093802
Title: Endoscopic Classification of Airway Obstruction and Drug Induced Sleep Endoscopy-Guided Surgery in Children With Obstructive Sleep-Disordered Breathing.
Brief Title: Endoscopic Classification and DISE-Guided Surgery in Pediatric Obstructive Sleep-Disordered Breathing.
Acronym: DISE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Hospital West Jutland (Other)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Mascha Eva Hildebrandt, MD, Regional Hospital West Jutland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: MHildebrandt
Record Dates: First submitted 2023-10-11; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Obstructive Sleep Apnea of Child
Keywords: Drug-induced Sleep Endoscopy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DISE-guided treatment group (Experimental): DISE findings will be documented and obstruction scored per pediatric DISE criteria. Clinically relevant obstruction is defined as >50% at minimum one site. (Adeno-)tonsillotomy will be performed if corroborative DISE suggests tonsil/adenoid obstruction; if not, no surgery will be performed.
  This approach is maintained despite other identified obstruction sites, which will be assessed at a later stage.
  Interventions: Diagnostic Test: Drug-induced Sleep Endoscopy findings (identified obstruction sites)
- Non-DISE-guided treatment group (Active Comparator): DISE findings will be documented, and video material will be saved for later assessment.
  Patients will be operated according to current guidelines (s.o.), regardless of perioperative DISE findings, i.e. tonsillotomy +/- adenoidectomy.
  Interventions: Diagnostic Test: Drug-induced Sleep Endoscopy findings (identified obstruction sites)

INTERVENTIONS:
Diagnostic Test: Drug-induced Sleep Endoscopy findings (identified obstruction sites) — As described above
  Other Names: Turbinoplasty; Nasal steroids

SUMMARY:
Pediatric obstructive sleep apnea (OSA) can lead to severe health issues if untreated. While polysomnography is the gold standard for diagnosis, current surgical treatment in Denmark relies on caregiver reports and clinical exams. Approximately 25% of patients have persistent symptoms post-surgery, indicating the need for better diagnostic and treatment options. Drug-Induced Sleep Endoscopy (DISE) allows dynamic upper airway visualization during mild sedation, aiding in treatment decisions. This research project aims to evaluate the impact of DISE-guided interventions on pediatric OSA outcomes and compare its effectiveness and cost/benefit with traditional diagnostic approaches.

DETAILED DESCRIPTION:
Background

1.1 Pediatric Obstructive Sleep Apnea

Pediatric OSA ranges from simple snoring to severe upper airway obstruction during sleep. Left untreated, it can lead to significant health issues, especially in children, impacting their cognitive development, learning, and social interactions.

1.2 Diagnostics and Surgical Strategies

Polysomnography (PSG) is the gold standard for diagnosing OSA. In Denmark, PSG isn't widely used due to equipment and setup constraints.

Surgical treatment for pediatric OSA in Denmark relies primarily on clinical examination of the tonsils and parental reports of symptoms.

1.3 Drug-Induced Sleep Endoscopy (DISE)

DISE is a method for visualizing upper airway collapse during sleep using a flexible endoscope. It is increasingly used to guide surgical decisions for pediatric OSA in various countries, though its clinical impact remains uncertain.

2. Aims

This research project aims to evaluate the impact of DISE-guided surgical interventions on pediatric OSA outcomes and compare the effectiveness of a DISE-inclusive diagnostic approach with the traditional pediatric OSA workup. The specific objectives are:

Evaluate treatment outcomes, including the reduction in persistent OSA post-surgery.

Classify and compare patterns of airway obstruction observed during DISE in surgically naive children.

Compare diagnostic approaches in terms of cost, time, and benefits. Identify adverse events and complications related to sedation and surgery. Assess the feasibility of DISE in Danish patients through a pilot study.

3. Methods

3.1 Randomized Controlled Trial (RCT)

Patients undergo initial clinical examination and home respiratory polygraphy (HRP). Based on AAO-HNSF criteria, patients with OSA will undergo DISE. The sample size for the RCT is 250 patients, with 125 in each group.

3.2 Statistics

Statistical analysis will involve Chi-square tests, logistic regression, and T-tests for comparisons between groups.

3.3 Sedation Protocol

Sedation will use propofol to induce a state similar to natural sleep, guided by preoperative polysomnography.

3.4 Assessment of Obstruction

Obstruction characteristics will be documented using the International Pediatric Sleep Endoscopy Scale (IPSES).

3.5 Follow-up

Patients will have two follow-up appointments at three and 12 months postoperatively, including clinical examination, HRP, and re-DISE at three months for both groups.

4. Outcomes

4.1 Primary Outcome

The primary outcome is the treatment failure rate, comparing the proportion of patients with persistent OSA post-surgery in the DISE-guided surgery group to the non-DISE-guided surgery group.

4.2 Secondary Outcomes

Secondary outcomes include evaluation of DISE findings, changes in apnea-hypopnea index (AHI), quality of life improvement, DISE-score/airway obstruction pattern, and identification of adverse events and complications.

4.3 Confounding Factors

Population characteristics, such as age, obesity (BMI), and gender, will be considered.

5. Ethical Considerations

In cases where no obstruction is identified related to tonsils or adenoids, alternative treatment options will be discussed with parents. Privacy and informed consent are required. The study will follow ethical and data protection regulations

ELIGIBILITY:
Inclusion Criteria:

* Surgically naïve, otherwise healthy, non-syndromic children aged 2-12 years with suspected oSDB of any severity
* One completed Pediatric Sleep Questionnaire - Sleep Related Breathing Disorder (PSQ)
* Home Respiratory Polygraphy (HRP) and/or in-house Polysomnography (PSG) showing OSA according to the definition of AAO-HNSF

Exclusion Criteria:

* Syndromes and congenital/acquired craniofacial abnormalities/malformations of the upper airways
* Neurological conditions affecting upper airway muscle tone
* Lower airway disease (tracheomalacia, asthma)
* Previous surgery of the nose/pharynx/larynx

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Failure Rate | one year post surgery
  Proportion of patients, who exhibit persistent OSA post-surgery in the DISE-guided surgery group compared to the non-DISE-guided surgery group (controls).

SECONDARY OUTCOMES:
DISE findings | initial assessment and one year post surgery
  Evaluation of DISE findings and pediatric VOTE:
  Assessing obstruction degree and sites in both groups.
  Quality of Life Improvement:
  DISE-score and Airway Obstruction Pattern:
  Identifying and comparing anatomical obstruction sites and severity during DISE in both groups.
OSA (AHI) | initial assessment and one year post surgery
  Change in apnea-hypopnea index (AHI):
  Analyzing AHI and oxygen saturation differences between baseline and post-treatment in both groups.
Quality of Life (OSA-18) | initial assessment and one year post surgery
  Evaluation of symptom changes and quality of life using the OSA-18 questionnaire in both groups.
Sedation-related and surgical complications | initial assessment and one year post surgery
  Adverse Events and Complications:
  Investigation of the incidence and severity of sedation-related events and surgical complications in both groups, including postoperative hemorrhage, infection, recurrent symptoms post-tonsillotomy, and symptom improvement without treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Therese E Ovesen, Prof. DMSc, Study Director — Regional Hospital West Jutland
Locations (1):
- Regional Hospital Gødstrup, Herning, Region of Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided